CLINICAL TRIAL: NCT01441791
Title: Protective Ventilation During General Anesthesia for Open Abdominal Surgery - a Randomized Controlled Trial
Brief Title: PROVHILO:Protective Ventilation During General Anesthesia for Open Abdominal Surgery
Acronym: PROVHILO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Principal Investigator and Clinical Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROVHILO; ISRCTN70332574 (Registry Identifier: Controlled Trials); NTR(TC=2517) (Registry Identifier: Dutch Trial Register); NCT01585116 (obsolete NCT alias)
Record Dates: First submitted 2011-09-23; First posted 2011-09-28 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Postoperative Respiratory Complications
Keywords: PEEP; Positive end-expiratory pressure; Recruitment maneuver; Open lung approach; Post-operative complications; Open abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lung protective strategy ventilation (Experimental): Lung protective strategy ventilation: PEEP at 12 cmH2O, Recruitment maneuvers (after intubation, after any disconnection from the mechanical ventilator, directly before detubation)
  Interventions: Procedure: Lung protective strategy ventilation
- Conventional Strategy (No Intervention): * PEEP at maximum 2 cmH2O, if possible 0 cmH2O
  * No recruitment maneuvers Patients are randomized and intra-operatively ventilated with conventional strategy (PEEP at maximum 2 cmH2O without recruitment maneuvers).

INTERVENTIONS:
Procedure: Lung protective strategy ventilation — Patients are randomized and intra-operatively ventilated with a lung protective strategy (PEEP at 12 cmH2O with recruitment maneuvers)
  Arms: Lung protective strategy ventilation

SUMMARY:
The purpose of this international, multicentre, double-blinded randomized controlled trial is to determine if the "open lung approach" providing recruitment maneuvers and PEEP(Positive End Expiratory Pressure) during general anesthesia reduces atelectasis formation and improves respiratory function in the immediate post-operative period after major abdominal surgery.

Participating centres throughout the world will include a total of 900 adult patients undergoing general anesthesia for open abdominal surgery with high or intermediate risk for post-operative pulmonary complications. Patients are randomized and intra-operatively ventilated with either a lung protective strategy (PEEP at 12 cmH2O with recruitment maneuvers) or a conventional strategy (PEEP at maximum 2 cmH2O without recruitment maneuvers). Patients will be assessed on the first 5 post-operative days, on day of discharge and on day 90 post-operative. Primary endpoint is any post-operative pulmonary complication (see below). Secondary endpoints are post-operative extra-pulmonary complications, intra-operative mechanical ventilation related complications, unscheduled ICU (Intensive Care Unit) (re-) admission, and length of hospital stay.

DETAILED DESCRIPTION:
Research questions

1. Does mechanical ventilation with the use of higher levels of PEEP(Positive End Expiratory Pressure) and intra-operative RMs (Recruitment maneuvers) protect against pulmonary complications in patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?
2. Does mechanical ventilation with the use of higher levels of PEEP and intra-operative RMs protect against extra-pulmonary complications in patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?
3. Does mechanical ventilation with the use of higher levels of PEEP and intra-operative RMs shorten length of hospital stay of patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?
4. Does mechanical ventilation with the use of higher levels of PEEP and intra-operative RMs ameliorate post-operative wound healing in patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?
5. Does mechanical ventilation with the use of higher levels of PEEP and intra-operative RMs attenuate post-operative unexpected need for ICU admission (i.e., before surgery the patient is not scheduled for admission to the ICU, but eventually is admitted) or ICU readmission in patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?
6. Does mechanical ventilation with the use of higher levels of PEEP and intra-operative RMs influence intra-operative complications related to the ventilator strategy (i.e., de-saturation, hypotension during recruitment, need for vasopressors) or ICU readmission in patients at high or intermediate risk for postoperative pulmonary complications scheduled for non-laparoscopic abdominal surgery?

Methods In this international randomized controlled trial all patients with high or intermediate risk for post-operative pulmonary complications following non-laparoscopic abdominal surgery with general anesthesia are eligible for participation. To identify such patients the ARISCAT risk score is used.

Patients are randomly assigned to mechanical ventilation with levels of PEEP at 12 cmH2O with the use of recruitment maneuvers (the lung-protective strategy) or mechanical ventilation with levels of PEEP at maximum 2 cmH2O without recruitment maneuvers (the conventional strategy).

Patients are ventilated with a volume-controlled mechanical ventilation strategy. Although it is left to the discretion of the attending anesthesiologist to use different fractions of inspired oxygen, it is advised to use at least 0.4, with the lowest oxygen fraction to maintain oxygen saturation ≥ 92%. The I:E ratio is set at 1:2, and the respiratory rate is adjusted to reach normocapnia (etCO2 between 35 and 45 mmHg). Tidal volumes of < 8 mL/kg predicted body weight (PBW) are advised to be used.

Recruitment maneuvers, as part of the lung-protective strategy, are performed directly after intubation, after any disconnection from the mechanical ventilator, and directly before tracheal extubation. Recruitment maneuvers should not be performed when patients are hemodynamic unstable, as judged by the attending physician. To obtain standardization among centers, recruitment maneuvers are performed as follows:

1. peak inspiratory pressure limit is set at 45 cmH2O
2. tidal volume is set at 8 ml/kg PBW and respiratory rate at 6-8 breaths/min (or lowest respiratory rate that anesthesia ventilator allows), while PEEP is set at 12 cmH2O
3. inspiratory to expiratory ratio (I:E) is set at 1:2
4. tidal volumes are increased in steps of 4 ml/kg PBW until a plateau pressure of 30-35 cmH2O
5. 3 breaths are administered with a plateau pressure of 30-35 cmH2O
6. peak inspiratory pressure limit, respiratory rate, I:E, and tidal volume are set back to settings preceding each recruitment maneuver, while maintaining PEEP at 12 cmH2O

The study protocol stresses that routine general anesthesia, post-operative pain management, physiotherapeutic procedures and fluid management must be used in the peri-operative as well as the post-operative period according to each centers specific expertise and routine clinical use, to minimize interference with the trial intervention.

Centres The investigators aim to recruit as many centres as possible worldwide, but expect a minimum of 40 centres.

Ethics approval National co-ordinators will be responsible for clarifying the need for ethics approval and applying for this where appropriate according to local policy. Centres will not be permitted to record data unless ethics approval or an equivalent waiver is in place. The investigators expect that in most, if not every participating country, a patient informed consent will be required.

Monitoring Monitoring of patient safety and reviewing of safety issues is performed by a designated independent Data Safety and Monitoring Board. The DSMB watches over the ethics of conducting the study in accordance with the Declaration of Helsinki. All (serious) adverse events will be collected by the National Coordinators and sent in a blinded fashion to a designated SAE manager, who presents the events to the DSMB for evaluation.

Interim analysis One main concern is not to withhold positive effects of the open lung mechanical ventilation strategy to the control group. Therefore, interim analyses are performed after 300 and 600 patients. The first interim analysis is performed when 300 patients have successfully been included and followed-up. If the intervention has a strong trend for improving post-operative pulmonary complications (as defined above) with a p-value < 0.0005 is found at 300 patients or < 0.014 at 600 patients, termination of the study is considered. The third and final analysis is performed at 900 patients with a p-value of 0.045 for significance. When post-operative pulmonary complications occur significantly more frequent in the intervention group, terminating the study due to harm will be considered when p ≤ 0.022 for each interim analysis.

Blinding The patient is blinded for the allocated treatment during the trial. In the participating centers at least 2 investigators are involved with the study. One researcher is involved with mechanical ventilation practice in the operation room, he/she will be blinded for the randomized intervention most closely to the time of tracheal intubation (depending on local situation) - the second investigator, blinded for randomization arm, will score the primary and secondary post-operative endpoints.

Data collection Data will be collected at inclusion pre-operatively, intra-operatively and post-operatively on day 1, day 2, day 3, day 4, day 5, day of discharge and on day 90. Data collection will be performed by an investigator blinded for the randomization group at the bedside, except on day 90 if the patient is discharged. In that case follow-up will be performed by telephone. Data will be coded by a patient identification number (PIN) of which the code will be kept safe at the local sites. The data will be transcribed by local investigators onto an internet based electronic CRF.

Sample size calculation The required sample size is calculated from an estimated effect size derived from data collected in the ARISCAT study and previous studies on the incidence of postoperative pulmonary complications. A two group χ2 test with a 0.05 two-sided significance level will have 80% power to detect the difference (in post-operative pulmonary complications) between conventional mechanical ventilation (24%) and open lung mechanical ventilation (16.5%) (Odds ratio of 0.626) when the sample size in each group is 450.

Statistical analysis Normally distributed variables will be expressed by their mean and standard deviation; not normally distributed variables will be expressed by their medians and interquartile ranges; categorical variables will be expressed as n (%). In test groups of continuous normally distributed variables, Student's t-test will be used. Likewise if continuous data are not normally distributed the Mann-Whitney U test will be used. Categorical variables will be compared with the Chi-square test or Fisher's exact tests or when appropriate as relative risks. Where appropriate statistical uncertainty will be expressed by 95% confidence levels.

Primary outcome is the total occurrence of pulmonary complications within the first 5 post-operative days, presented as a percentage. The percentage will be analyzed as continuous data. If the data is normally distributed, Student's t-test will be used or when not normally distributed the Mann-Whitney U test will be used.

As this is a randomized controlled trial, we expect that randomization in this large study population will sufficiently balance the baseline characteristics. Baseline balance is tested and imbalance compensated in all pre-operative variables and on ARISCAT scores. However if imbalance occurs, the confounding factor will be corrected using a multiple logistic regression model. For this we will treat the proportion as a binary response (complications occur during day one to day five post-operative).

Time to event variables (primary and secondary outcomes) are analyzed using a proportional hazard model adjusted for possible imbalances of patients' baseline characteristics. Time course variables (e.g. repeated measures of vital parameters, blood values, VAS-scores, actual mobility) are analyzed by a linear mixed model. The linear mixed models procedure expands the GLM so that the data are permitted to exhibit correlated and non-constant variability. The model includes two factors: 1) study group (fixed factor, intervention or control group), each level of the study group factor can have a different linear effect on the value of the dependent variable; 2) time as a covariate, time is considered to be a random sample from a larger population of values, the effect is not limited to the chosen times.

Organization The study is conducted by the PROVHILO collaboration. National co-ordinators will lead the project within individual nations and identify participating hospitals, translate study paperwork, distribute study paperwork and ensure necessary regulatory approvals are in place. They provide assistance to the participating clinical sites in trial management, record keeping and data management. Local coordinators in each site will perform randomization and mechanical ventilation, supervise data collection and ensure adherence to Good Clinical Practice during the trial.

Study Population Adult patients with high or intermediate risk for postoperative pulmonary complications undergoing open abdominal surgery with general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Open abdominal surgery
* General anesthesia
* High or intermediate risk for postoperative pulmonary complications according to ARISCAT score [J.Canet et al, Anesthesiology 2010;113]

Exclusion Criteria:

* Age > 18 years
* Body mass index > 40 kg/m2
* Laparoscopic surgery
* Previous lung surgery (any)
* Persistent hemodynamic instability, intractable shock (considered hemodynamic unsuitable for the study by the patient's managing physician)
* History of previous severe chronic obstructive pulmonary disease (COPD) (non-invasive ventilation and/or oxygen therapy at home, repeated systemic corticosteroid therapy for acute exacerbations of COPD)
* Recent immunosuppressive medication (receiving chemotherapy or radiation therapy within last 2 months)
* Severe cardiac disease (New York Heart Association class III or IV, or acute coronary syndrome, or persistent ventricular tachyarrhythmia's)
* Mechanical ventilation > than 30 minutes (e.g., in cases of general anesthesia because of surgery) within last 30 days
* Pregnancy (excluded by laboratory analysis)
* Acute lung injury or acute respiratory distress syndrome expected to require prolonged postoperative mechanical ventilation
* Neuromuscular disease (any)
* Consented for another interventional study or refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Post-operative pulmonary complications (PPCs) | first 5 days post-operative and on the day of discharge a final assessment is performed scoring endpoints occuring on day 6 and up.
  Mild respiratory failure Severe respiratory failure ALI/ARDS (Acute Lung Injury and Acute Respiratory Distress Syndrome) Suspected pulmonary infection Pulmonary infiltrate Pleural effusion Atelectasis Pneumothorax Bronchospasm Aspiration pneumonitis Cardiopulmonary edema

SECONDARY OUTCOMES:
Post-operative extra-pulmonary complications | first 5 days post-operative and on the day of discharge a final assessment is performed scoring endpoints occuring on day 6 and up
Intra-operative mechanical ventilation related complications | during the length of anesthesia, which will be an estimated 2 to 5 hours
Unscheduled Intensive Care Unit (ICU) (re-) admission | first 5 days post-operative and on the day of discharge a final assessment is performed scoring endpoints occuring on day 6 and up
Length of hospital stay on day 90 | until day 90 post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD, Principal Investigator — Department of Intensive Care, Academic Medical Center, University of Amsterdam; Paolo Pelosi, MD, Principal Investigator — Department of Surgical Sciences and Integrated Diagnostics, University of Genoa, Italy; Marcelo Gama de Abreu, MD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, University Hospital Carl Gustav Carus, Technical University Dresden, Germany; Sabrine NT Hemmes, MD, Study Director — PROVHILO Study Trial Coordinator, Department of Intensive Care and Anesthesiology, Academic Medical Center, University of Amsterdam, The Netherlands
Locations (30):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinics, Rochester, New York
- Medical University,, Vienna, Austria
- Belgium (4):
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - AZ Sint-Jan, Bruges
  - UZ Gent, Ghent
  - Virga Jesse Hospital, Hasselt
- Hospital Clínico de la Pontificia Universidad Católica de Chile, Santiago, Chile, Santiago, Chile
- University Hospital Sveti Duh, Zagreb, Croatia
- Germany (5):
  - University Hospital of Bonn Medical School, Bonn
  - University Clinic Carl Gustav Carus, Dresden, Germany, Dresden
  - Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - University of Leipzig, Leipzig
  - University Medical Center Mainz, Mainz
- Italy (9):
  - Università degli Studi di Catanzaro, Catanzaro
  - University of Foggia, Foggia
  - Università degli Studi di Genova, Genoa
  - Università degli Studi di Napoli Federico II , Napoli, Italy, Napoli
  - Università degli Studi di Palermo, Palermo
  - Università degli Studi di Roma Cattolica, Rome
  - Hospital of Rivoli, Turin
  - Università degli Studi di Udine, Udine
  - Università degli Studi dell'Insubria, Varese
- Academic Medical Centre, Amsterdam, Netherlands
- Spain (4):
  - Fundació Puigvert (IUNA), Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Germans Trias I Pujol, Barcelona, Spain, Barcelona
  - Consorcio Hospital General Universitario de Valencia, Valencia
- United Kingdom (2):
  - Barts Health NHS Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- [Background] Hemmes SN, Severgnini P, Jaber S, Canet J, Wrigge H, Hiesmayr M, Tschernko EM, Hollmann MW, Binnekade JM, Hedenstierna G, Putensen C, de Abreu MG, Pelosi P, Schultz MJ. Rationale and study design of PROVHILO - a worldwide multicenter randomized controlled trial on protective ventilation during general anesthesia for open abdominal surgery. Trials. 2011 May 6;12:111. doi: 10.1186/1745-6215-12-111. PMID 21548927
- [Background] J. Canet et al, Anesthesiology 2010;113 http://www.ncbi.nlm.nih.gov/pubmed/21045639
- [Derived] Serpa Neto A, Bos LD, Campos PPZA, Hemmes SNT, Bluth T, Calfee CS, Ferner M, Guldner A, Hollmann MW, India I, Kiss T, Laufenberg-Feldmann R, Sprung J, Sulemanji D, Unzueta C, Vidal Melo MF, Weingarten TN, Tuip-de Boer AM, Pelosi P, Gama de Abreu M, Schultz MJ; PROVHILO* and the PROVE** investigators. Association between pre-operative biological phenotypes and postoperative pulmonary complications: An unbiased cluster analysis. Eur J Anaesthesiol. 2018 Sep;35(9):702-709. doi: 10.1097/EJA.0000000000000846. PMID 29957706
- [Derived] Treschan TA, Schaefer M, Kemper J, Bastin B, Kienbaum P, Pannen B, Hemmes SN, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Ventilation with high versus low peep levels during general anaesthesia for open abdominal surgery does not affect postoperative spirometry: A randomised clinical trial. Eur J Anaesthesiol. 2017 Aug;34(8):534-543. doi: 10.1097/EJA.0000000000000626. PMID 28306591
- [Derived] Serpa Neto A, Campos PP, Hemmes SN, Bos LD, Bluth T, Ferner M, Guldner A, Hollmann MW, India I, Kiss T, Laufenberg-Feldmann R, Sprung J, Sulemanji D, Unzueta C, Melo MF, Weingarten TN, Boer AM, Pelosi P, Gama de Abreu M, Schultz MJ; PROVE Network Investigators. Kinetics of plasma biomarkers of inflammation and lung injury in surgical patients with or without postoperative pulmonary complications. Eur J Anaesthesiol. 2017 Apr;34(4):229-238. doi: 10.1097/EJA.0000000000000614. PMID 28187051
- See also: PROVHILO website — https://sites.google.com/site/provhilo/